CLINICAL TRIAL: NCT05975762
Title: Outcome of Surgical Fixation of Multiple Fractured Ribs at Sohag University Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hossam Hassan Sayed, resident at cardiothoracic department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-07-09MS
Record Dates: First submitted 2023-07-24; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Multiple Fractures of Ribs
MeSH Terms: interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): surgical fixation group
  Interventions: Procedure: surgical rib fixation
- control group (No Intervention): conservation group

INTERVENTIONS:
Procedure: surgical rib fixation — open reduction and internal rib fixation
  Other Names: open reduction and internal fixation
  Arms: intervention group

SUMMARY:
The ribs are rigid and flexible structures that make up the chest skeleton and are a set of twelve paired bones. After Blunt trauma rib fractures incidence is about 30 to 40% [1].

Due to trauma, (4th -9th) ribs are often affected and the fracture point of the ribs is often on the midaxillary line. In ( 1st&2nd) ribs fractures subclavian vessels and brachial plexus damage may occur. In fractures in the lower ribs (8th-12th ribs), intra-abdominal organs injury such as liver, spleen and kidney should be investigated. 11-12. ribs fractures are rare because the ribs are more flexible (floating).

Pain is the most important symptom indicating rib fracture, and it usually increases with coughing, breathing, and movement. Broken rib ends can be felt with palpation with sever tenderness at the site of fracture. Pneumothorax and/or hemothorax may develop as a result of the sharp end of the broken rib causing lung parenchymal damage[2].

ELIGIBILITY:
Inclusion Criteria:

* multiple fractured ribs pre ventilation

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
mechanical ventilation | 1 year
  the need and duration of mechanical ventilation
thoracic pain | 1 year
  measure severity of pain using pain scale 0 to10.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marasco SF, Martin K, Niggemeyer L, Summerhayes R, Fitzgerald M, Bailey M. Impact of rib fixation on quality of life after major trauma with multiple rib fractures. Injury. 2019 Jan;50(1):119-124. doi: 10.1016/j.injury.2018.11.005. Epub 2018 Nov 3. PMID 30442372
- [Background] Schuurmans J, Goslings JC, Schepers T. Operative management versus non-operative management of rib fractures in flail chest injuries: a systematic review. Eur J Trauma Emerg Surg. 2017 Apr;43(2):163-168. doi: 10.1007/s00068-016-0721-2. Epub 2016 Aug 29. PMID 27572897
- [Background] Beks RB, Peek J, de Jong MB, Wessem KJP, Oner CF, Hietbrink F, Leenen LPH, Groenwold RHH, Houwert RM. Fixation of flail chest or multiple rib fractures: current evidence and how to proceed. A systematic review and meta-analysis. Eur J Trauma Emerg Surg. 2019 Aug;45(4):631-644. doi: 10.1007/s00068-018-1020-x. Epub 2018 Oct 1. PMID 30276722